CLINICAL TRIAL: NCT00183794
Title: Phase II Clinical Trial of Docetaxel in Combination With Gemcitabine in Platinum-Resistant Ovarian Cancer and Primary Peritoneal Carcinoma
Brief Title: Clinical Trial of Docetaxel in Combination With Gemcitabine in Platinum-Resistant Ovarian Cancer and Primary Peritoneal Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Aventis Pharmaceuticals (Industry); Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5GYN-02-2
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Results first posted 2013-01-25 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2012-12

CONDITIONS: Ovarian Carcinoma; Peritoneal Neoplasms
Keywords: Primary Peritoneal
MeSH Terms: conditions — Ovarian Neoplasms; Peritoneal Neoplasms | interventions — Docetaxel; Gemcitabine

ARMS (1):
- Arm 1 (Experimental): Patients will receive Docetaxel 75mg/m2 IV over 15-30 minutes on day 1 followed by Gemcitabine 800 mg/m2 IV over 30 minutes on Days 1 and 8. Cycles will be repeated every 3 weeks.
  Interventions: Drug: Docetaxel and Gemcitabine

INTERVENTIONS:
Drug: Docetaxel and Gemcitabine — Docetaxel 75 mg/m2 IV over 15-30 minutes on day 1 followed by Gemcitabine 800 mg/m2 IV over 30 minutes on Days 1 and 8 of each 3 weeks (21 days) cycle.

SUMMARY:
This study is for patients with advanced ovarian cancer that has reappeared after treatment with conventional therapy. The purpose of this study is to determine if the combination of docetaxel and gemcitabine will be effective in reducing or eliminating the tumor(s) in patients with ovarian cancer.

Docetaxel is approved by the Food and Drug Administration (FDA) for the treatment of breast and lung cancer; gemcitabine is approved by the FDA for the treatment of pancreatic and lung cancer. Neither docetaxel nor gemcitabine are approved for the treatment of ovarian cancer. Both drugs have been shown to decrease the size of ovarian cancer tumors.

DETAILED DESCRIPTION:
Primary Objective:

1. To determine the response rate, time to progression and survival (secondary) of the combination of docetaxel and gemcitabine administered on a weekly basis to patients with platinum-resistant ovarian cancer

Secondary Objective:

1. To determine the toxicity of this combination regimen in patients with platinum-resistant ovarian cancer
2. To evaluate the toxicity and safety profile of a short course (one dose) of premedication with steroids to patients receiving weekly gemcitabine and docetaxel

OUTLINE: Patients receive gemcitabine IV over 30 minutes on days 1 and 8, and docetaxel IV over 60 minutes on day 8. Treatment repeats every 21 days until PD, unacceptable toxicity, or patient's withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven diagnosis of epithelial ovarian ca
* Must have platinum-resistant disease. (Defined as progression during the most recent platinum-based chemotx or relapse < 6 months after the most recent platinum-based chemotx regimen.)
* Measurable or evaluable disease. (Patients whose dz is manifested only as an elevated CA-125 [greater than or equal to 100] are eligible. If an elevated CA-125 is the only manifestation of dz, it must be confirmed on 2 separate times, at least 2 weeks apart. Patients with positive cytology only are not eligible.)
* Greater than or equal to 18 years of age
* GOG performance status less than or equal to 2
* AGC/ANC greater than or equal to 1.5; platelets greater than or equal to 100,000; hemoglobin (Hgb) greater than or equal to 8.0.
* Creatinine less than or equal to 2.0
* Total bilirubin less than or equal to upper limit of normal (uln)
* SGOT and/or SGPT less than or equal to 2.5 x uln if alkaline phosphatase less than or equal to uln, or alkaline phosphatase less than or equal to 4 x uln if transaminases are less than or equal to uln. (If both SGOT/SGPT >1.5 x uln and alkaline phosphatase > 2.5 x uln, patient is not eligible.)
* Fully recovered from acute toxicities secondary to prior treatment (tx)
* Signed informed consent

Exclusion Criteria:

* Prior treatment with gemcitabine or docetaxel
* Underlying medical, psychiatric, or social conditions that would preclude patient from receiving treatment
* Peripheral neuropathy greater than or equal to Grade 2
* No prior tx with cisplatin or carboplatin

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2002-11; Primary Completion 2009-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Agustin Garcia, MD, Principal Investigator — University of Southern California
Locations (1):
- Norris Comprehensive Cancer Center, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the USC+LAC Women's Hospital and the USC/Norris Cancer Hospital between December 2002 and April 2008.
Groups:
- Gemcitabine and Docetaxel: Patients will receive Docetaxel 75mg/m2 IV over 15-30 minutes on day 1 followed by Gemcitabine 800 mg/m2 IV over 30 minutes on Days 1 and 8. Cycles will be repeated every 3 weeks.
Period: Overall Study
Arm/Group | Gemcitabine and Docetaxel
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Gemcitabine and Docetaxel
Number analyzed (Participants) | 20
Age, Continuous [Median (Full Range); unit: years]
  Between 43 and 75 years | 59 [43 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 12
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response Type: CR, PR, SD or PD
Description: Tumor response will be based on the RECIST v1.0 criteria. CR (complete response)= disappearance of all target lesions, PR (partial response)= greater or equal to 30% decrease in sum of longest diameter of target lesions, SD (stable disease)= <30% decrease or <20% increase, PD (progressive disease)= greater or equal to 20% increase in longest diameter of target lesions. For patients with an elevated CA-125 as the only evidence of disease, a PR was defined as a decrease of 50% or more lasting at least 8 weeks (Rustin et al. JCO 14:1545-51, 1996). Disease assessment performed every 2 cycles (1 cycle = 21 days). Responders included CR and PR.
Time Frame: 6 months after enrollment of last participant
Population: Participants with evaluable or measurable tumor, who complete 2 courses of treatment will be included in analysis of tumor response.
Measure: Number; unit: Participants
Arm/Group | Gemcitabine and Docetaxel
Number analyzed (Participants) | 20
Participants
  CR | 1 [0.087 to 0.49]
  PR | 4
  SD | 9
  PD | 6

2. Secondary Outcome: Median Time to Progression (Months)
Description: Defined as the time from first day of treatment to the first observation of disease progression or death due to any cause. If a patient has not progressed or died, progression-free survival is censored at the time of last follow-up. Progression based on RECIST v1.0 criteria for measurable disease, and on CA-125 for patients with an elevated CA-125 as the only evidence of disease (Rustin et al. JCO 14:1545-51, 1996)
Time Frame: 6 months after enrollment of last patient
Population: All participants who receive the first course of treatment are included in the summary of PFS.
Measure: Median (Full Range); unit: Months
Arm/Group | Gemcitabine and Docetaxel
Number analyzed (Participants) | 20
Months | 3 [1 to 23]

ADVERSE EVENTS:
Arm/Group | Gemcitabine and Docetaxel
Serious Adverse Events (participants affected / at risk) | 12/20
Other Adverse Events (participants affected / at risk) | 13/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine and Docetaxel (N=20)
Alkaline Phosphatase Increased (Investigations) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Neutrophil Count Decreased (Investigations) | 11 (29)
Platelet Count Decreased (Investigations) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
White Blood Cell Decreased (Investigations) | 5 (12)
Wound Infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine and Docetaxel (N=20)
Nausea (Gastrointestinal disorders) | 4 (4)
Peripheral Motor Neuropathy (Nervous system disorders) | 2 (2)
Fatigue (General disorders) | 7 (12)
Creatinine Increased (Investigations) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (13)
Neutrophil Count Decreased (Investigations) | 1 (12)
White Blood Cell Decreased (Investigations) | 10 (14)
Vomiting (Gastrointestinal disorders) | 2 (2)
Ascites (Gastrointestinal disorders) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Peripheral Sensory Neuropathy (Nervous system disorders) | 6 (9)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Palpitations (Cardiac disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (5)
Pin (General disorders) | 1 (1)
Rash/Acneiform (Skin and subcutaneous tissue disorders) | 4 (7)
Platelet Count Decreased (Investigations) | 7 (13)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Blood Bilirubin Increased (Investigations) | 1 (1)
Alkaline Phosphatase (Investigations) | 3 (3)
Constipation (Gastrointestinal disorders) | 3 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (5)
Localized Edema (General disorders) | 4 (6)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (2)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Dizziness (Nervous system disorders) | 3 (4)
Skin Disorder - Other (specify: skin tear) (Skin and subcutaneous tissue disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 2 (3)
Nail Discoloration (Skin and subcutaneous tissue disorders) | 3 (3)
Bruising (Injury, poisoning and procedural complications) | 2 (2)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1)
Fever (General disorders) | 3 (5)
Weight Gain (Investigations) | 1 (2)
Aspartate Aminotrasferase Increased (Investigations) | 3 (5)
Alanine Aminotransferase Increased (Investigations) | 3 (5)
Chills (General disorders) | 3 (4)
Urinary Tract Pain (Renal and urinary disorders) | 1 (1)
Mucosits Oral (Gastrointestinal disorders) | 2 (4)
Watering Eyes (Eye disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Anorexia (Metabolism and nutrition disorders) | 2 (3)
Hot Flashes (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes